CLINICAL TRIAL: NCT01378676
Title: A Phase II, Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Effects of Multiple Doses of CK-2017357 in Patients With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: A Study to Evaluate the Effects of Multiple Doses of CK-2017357 in Patients With Amyotrophic Lateral Sclerosis (ALS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cytokinetics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CY 4024
Record Dates: First submitted 2011-06-20; First posted 2011-06-22 (Estimated); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — CK-2017357; Riluzole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Matching Placebo (Placebo Comparator)
  Interventions: Drug: Placebo (Part A); Drug: Riluzole 50 MG (Part B); Drug: Placebo (Part B)
- Active Drug Low Dose (CK-2017357 125 mg) (Experimental)
  Interventions: Drug: Placebo (Part A); Drug: CK-2017357 (Part A); Drug: Riluzole 50 MG (Part B); Drug: Placebo (Part B); Drug: CK-2017357 (Part B)
- Active Drug Mid Dose (CK-2017357 250 mg) (Experimental)
  Interventions: Drug: Placebo (Part A); Drug: CK-2017357 (Part A); Drug: Riluzole 50 MG (Part B); Drug: Placebo (Part B); Drug: CK-2017357 (Part B)
- Active Drug High Dose (CK-2017357 375 mg) (Experimental)
  Interventions: Drug: CK-2017357 (Part A); Drug: Riluzole 50 MG (Part B); Drug: CK-2017357 (Part B)

INTERVENTIONS:
Drug: Placebo (Part A) — Placebo tablets once daily for 14 days (Part A)
  Arms: Active Drug Low Dose (CK-2017357 125 mg); Active Drug Mid Dose (CK-2017357 250 mg); Matching Placebo
Drug: CK-2017357 (Part A) — One 125 mg CK-2017357 tablet once daily for 14 days (Part A)
  Other Names: tirasemtiv
  Arms: Active Drug Low Dose (CK-2017357 125 mg)
Drug: CK-2017357 (Part A) — Two 125 mg CK-2017357 tablets once daily for 14 days (Part A)
  Other Names: tirasemtiv
  Arms: Active Drug Mid Dose (CK-2017357 250 mg)
Drug: CK-2017357 (Part A) — Three 125 mg CK-2017357 tablets once daily for 14 days (Part A)
  Other Names: tirasemtiv
  Arms: Active Drug High Dose (CK-2017357 375 mg)
Drug: Riluzole 50 MG (Part B) — One 50 mg tablet once daily for 14 days (Part B)
Drug: Placebo (Part B) — Placebo tablets once daily for 14 days (Part B)
  Arms: Active Drug Low Dose (CK-2017357 125 mg); Active Drug Mid Dose (CK-2017357 250 mg); Matching Placebo
Drug: CK-2017357 (Part B) — One 125 mg tablet once daily for 14 days (Part B)
  Other Names: tirasemtiv
  Arms: Active Drug Low Dose (CK-2017357 125 mg)
Drug: CK-2017357 (Part B) — Two 125 mg tablets once daily for 14 days (Part B)
  Other Names: tirasemtiv
  Arms: Active Drug Mid Dose (CK-2017357 250 mg)
Drug: CK-2017357 (Part B) — Three 125 mg tablets once daily for 14 days (Part B)
  Other Names: tirasemtiv
  Arms: Active Drug High Dose (CK-2017357 375 mg)

SUMMARY:
The study will generate data on safety, tolerability and pharmacokinetics after multiple daily doses of CK-2017357 in patients with ALS. Patients will be randomized into one of four different treatment groups, receiving daily oral doses of either placebo, 125 mg, 250 mg, or 375 mg of CK-2017357 for 14 days.

DETAILED DESCRIPTION:
In Part A, approximately 24 patients will be randomized to one of four different treatment groups. After a 7-day washout of riluzole, patients in each treatment group will receive daily oral doses of placebo, 125 mg, 250 mg, or 375 mg of CK-2017357 for 14 days. Patients will take daily doses of CK-2017357 or placebo (Day 1 through Day 14) and will return to the study site on Day 2, Day 8 and Day 15. All patients will return for a follow-up visit 7 days (± 2 days) after their last dose.

In Part B, approximately additional 24 patients will be randomized to one of four different treatment groups as in Part A. Patients in Part B will be required to decrease their riluzole dose to 50 mg once a day (QD) for 7 days prior to randomization. After this 7 day period, patients will take riluzole at 50 mg QD concurrently with their morning dose of blinded study drug.

ELIGIBILITY:
Key Inclusion Criteria:

1. Able to comprehend and willing to sign an Informed Consent Form (ICF)
2. Males or females 18 years of age or older
3. A diagnosis of familial or sporadic ALS (defined as meeting the possible, laboratory-supported probable, probable, or definite criteria for a diagnosis of ALS according to the World Federation of Neurology El Escorial criteria)
4. Maximum voluntary grip strength in at least one hand between 10 & 40 pounds (females) and 10 & 60 pounds (males)
5. Upright Slow Vital Capacity (SVC) >50% of predicted for age, height, and sex
6. Able to swallow tablets with water
7. Willing and able to remain off riluzole for 4 weeks (Part A only)
8. Currently taking and tolerating a stable dose of 50 mg BID riluzole (Part B only)
9. Willing and able to reduce daily dose of riluzole to 50 mg for 4 weeks (Part B only)
10. Willing and able to refrain from caffeine-containing products during study participation
11. Willing and able to remain off warfarin and theophylline-containing medications during study participation
12. Has a caregiver who is capable of observing and reporting patient status, and also assisting in the proper use of nocturnal oximetry equipment
13. Able to perform pulmonary function tests

Key Exclusion Criteria:

1. Life expectancy <3 months
2. Participation in any trial in which receipt of investigational study drug occurred within 30 days or 5 half-lives of the prior agent, whichever is greater, prior to dosing
3. Any prior treatment with CK-2017357
4. Use of non-invasive positive pressure ventilation (NIPPV) for any part of the day or night

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2011-06; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 21 days
  Safety and tolerability of CK-2017357 after multiple oral doses to steady state in patients with ALS

SECONDARY OUTCOMES:
Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) | 21 days
  An instrument for evaluating the functional status of patients with ALS. Minimum score is 0 and maximum score is 40. The higher the score the more function is retained.
Measurement of Grip Strength and Handgrip Fatigue | 21 days
  Measured using the DynEx Electronic Hand Dynamometer. Patients asked to squeeze the device with the maximum possible force to establish the maximum voluntary contraction. Handgrip fatigue is then measured. Patient is asked to squeeze the device until they can no longer stay above 60% of target or 120 seconds.
Measurement of muscle strength | 21 days
  Muscle strength is measured using Hand Held Dynamometry. A series of assessments are done on different muscle groups.
Measurement of Slow Vital Capacity (SVC) | 21 days
  SVC will be measured using the ndd EasyOne Spirometer System at Screening, Day -7, Day 1, Day 2, Day 8, Day 15 and at the Follow-Up Visit
Measurement of Sniff Nasal Inspiratory Pressure (SNIP) | 21 days
  SNIP will be measured using the Micro Medical Respiratory Pressure Meter (MicroRPM) at Screening, Day -7, Day 1, Day 2, Day 8, Day 15 and at the Follow-Up Visit
Measurement of Maximum Voluntary Ventilation (MVV) | 21 days
  MVV will be measured using the EasyOne Spirometer System at Screening, Day -7, Day 1, Day 2, Day 8, Day 15 and at the Follow-Up Visit
Patient global assessment | 15 days
  Patients will be asked to assess whether they feel the same, better or worse as compared to how they felt at pre-dose on Day 1
Investigator global assessment | 15 days
  Investigator will assess whether the patient appears the same, better or worse as compared to the patient's status at pre-dose on Day 1.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Shefner, MD, PhD, Study Chair — State University of New York - Upstate Medical University
Locations (9):
- United States (9):
  - California Pacific Medical Center, San Francisco, California
  - Mayo Florida, Jacksonville, Florida
  - University of Kansas, Kansas City, Kansas
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Columbia University Medical Center, New York, New York
  - SUNY Upstate Medical Center, Syracuse, New York
  - Carolinas Neuromuscular ALS-MND Center, Charlotte, North Carolina
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Drexel University College of Medicine, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Shefner JM, Watson ML, Meng L, Wolff AA; Neals/Cytokinetics STUDY Team. A study to evaluate safety and tolerability of repeated doses of tirasemtiv in patients with amyotrophic lateral sclerosis. Amyotroph Lateral Scler Frontotemporal Degener. 2013 Dec;14(7-8):574-81. doi: 10.3109/21678421.2013.822517. Epub 2013 Aug 19. PMID 23952636